CLINICAL TRIAL: NCT04932941
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Proof-of-concept, Phase IIA Study of MP1032 Plus Standard of Care vs Standard of Care in the Treatment of Hospitalized Participants With Moderate to Severe COVID-19
Brief Title: MP1032 Treatment in Patients With Moderate to Severe COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MetrioPharm AG (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP1032-CT05; 2021-000344-21 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: COVID-19; MP1032
MeSH Terms: conditions — COVID-19 | interventions — sodium luminolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MP1032 (Experimental): Participants will receive MP1032 300 milligrams (mg) twice daily (BID) with hospital selected SoC for 28 days.
  Interventions: Drug: MP1032
- Placebo (Placebo Comparator): Participants will receive placebo matched to MP1032 with hospital selected SoC for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP1032 — Hard gelatin capsules for oral administration.
  Arms: MP1032
Drug: Placebo — Placebo capsules matched to MP1032 for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MP1032 with standard of care (SoC) verses placebo with SoC in hospitalized adults participants with moderate to severe coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is admitted to hospital and has a positive severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) test by standard reverse transcription-polymerase chain reaction (RT-PCR) assay or equivalent test
* Participant has the presence of any symptom(s) suggestive of moderate or severe systemic illness with COVID-19

Key Exclusion Criteria:

* Participant, in opinion of the investigator, is not likely to survive >=48 hours beyond Day 1
* Participant has a diagnosis of asymptomatic COVID-19, mild COVID-19, or critical COVID-19 on Day 1
* Participant has a documented medical history of infection with hepatitis A, B, C, or with human immunodeficiency virus (with a detectable viral load and CD4 count <500 cells per micro liter), or a documented active infection with tuberculosis.
* The Participant has clinically significant electrocardiogram (ECG) abnormalities at screening

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (2):
  - Snake River Research PLLC, Idaho Falls, Idaho
  - Richmond University Medical Center, Staten Island, New York
- Bulgaria (7):
  - MHAT Blagoevgrad AD, Blagoevgrad
  - MHAT Sv. Ivan Rilski Kozloduy, Kozloduy
  - MHAT Dr. Stamen Iliev AD, Montana
  - SHATPD Pernik EOOD, Pernik
  - MHAT Dr. Ivan Seliminski AD, Sliven
  - Umhatem"N.I.Pirogov", Sofia
  - SHATPPD Sata Zagora EOOD, Stara Zagora
- France (3):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CHU de Grenoble Alpes, Grenoble
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Hungary (2):
  - DE KK Infektológiai Klinika, Debrecen
  - Flor Ferenc Hospital of Pest County, Kistarcsa
- Italy (7):
  - Ospedale GB Morgagni, Forlì
  - Ospedale SM Goretti, Latina
  - ASST-FBF-SACCO - Ospedale Luigi Sacco, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Policlinico di Napoli, Napoli
  - Ospedale "Santo Spirito! Pescara, Pescara
  - Policlinico Agostino Gemelli, Roma
- Romania (4):
  - Spitalul Clinic de Boli Infectioase si Tropicale "Dr. Victor Babes", Bucharest
  - Spitalul Municipal Caracal, Caracal
  - Spitalul Clinic de Boli Infectioase "Sfanta Parascheva", Iași
  - Clinica Anestezie si Terapie Intensiva, Timișoara
- Spain (6):
  - Hospital Clinic de Barcelona Hospital Clinic i Provincial, Barcelona
  - Hospital Ramon y Cajal, Edificio Central, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla/IDIVAL, Santander
  - Hospital Universitario de Valme, Seville
  - Hospital Álvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 sites in 6 countries from 19 October 2021 to 05 September 2022. Participants were randomized in the 2:1 ratio to treatment groups using an Interactive Web Response System (IWRS).
Pre-assignment Details: A total of 134 participants were screened, of which 132 participants were randomized to either the MP1032 plus standard of care (SoC) group or the placebo plus SoC group.
Groups:
- MP1032 300mg + SoC: Participants received MP1032, 300 milligrams (mg) hard gelatin capsules orally, twice daily (BID) with hospital selected SoC procedure for 28 days.
- Placebo + SoC: Participants received placebo matched to MP1032 hard gelatin capsules orally, BID with hospital selected SoC procedure for 28 days.
Period: Overall Study
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Started | 87 | 45
Intention-to-Treat Set (ITT) (The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study.) | 87 | 45
Pharmacokinetic Analysis Set (The Pharmacokinetic Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose.) | 4 | 0
Safety Set (The Safety Set included all randomized participants who received at least 1 dose of study drug.) | 86 | 45
Completed | 73 | 38
Not Completed | 14 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study.
Groups:
- MP1032 300mg + SoC: Participants received MP1032, 300mg hard gelatin capsules orally, BID with hospital selected SoC procedure for 28 days.
- Total: Total of all reporting groups
Arm/Group | MP1032 300mg + SoC | Placebo + SoC | Total
Number analyzed (Participants) | 87 | 45 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.83) | 62.3 (14.15) | 60.5 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 19 | 55
  Male | 51 | 26 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 79 | 44 | 123
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 87 | 45 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression Using National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale at Day 14
Description: Disease progression was defined as the percentage of participants who were not alive or who had respiratory failure. Respiratory failure was defined as participants who had a score of 2, 3 or 4 on the NIAID 8-point ordinal scale: The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status.
Time Frame: At Day 14
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 82 | 43
percentage of participants | 9.8 [4.307 to 18.321] | 11.6 [3.885 to 25.083]
Statistical Analysis 1: Comparison: MP1032 300mg + SoC vs Placebo + SoC; Test type: Superiority; p = 0.962, Mantel Haenszel; Common risk difference = -0.276, 95% CI 2-sided [-11.634 to 11.081] — Strata-adjusted Mantel Haenszel (MH) method for difference in proportions controlling for stratification factors (COVID-19 severity: moderate, severe, and age group: less than or equal to 65 years, greater than 65 years)

2. Secondary Outcome: Percentage of Participants With Disease Progression Using NIAID 8-point Ordinal Scale at Day 28
Description: Disease progression was defined as the percentage of participants who were not alive or who had respiratory failure. Respiratory failure was defined as participants who had a score of 2, 3 or 4 on the NIAID 8-point ordinal scale: The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 79 | 41
percentage of participants | 2.5 [0.308 to 8.848] | 2.4 [0.062 to 12.855]

3. Secondary Outcome: Percentage of Participants With Disease Resolution at Day 28
Description: Disease resolution was defined as participants who were alive and had a score of 6, 7, or 8 on the NIAID 8-point ordinal scale. The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 79 | 41
percentage of participants | 97.5 [91.152 to 99.692] | 97.6 [87.145 to 99.938]

4. Secondary Outcome: All-cause Mortality Rate up to Day 28
Description: All-cause mortality rate was the percentage of participants in each treatment group who died by Day 28 were reported.
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 82 | 42
percentage of participants | 2.4 [0.297 to 8.534] | 2.4 [0.060 to 12.566]

5. Secondary Outcome: Change From Baseline in Clinical Status Score Related to COVID-19 According to the NIAID 8-point Ordinal Scale at Day 28
Description: The NIAID 8-point Ordinal Scale is an assessment of the clinical status on a given study day and the scale was defined as follows: 1=Death, 2=Hospitalized, on invasive ventilation (mechanical ventilator and/or ECMO), 3=Hospitalized, on non-invasive ventilation or high-flow oxygen devices, 4=Hospitalized, requiring supplemental oxygen, 5=Hospitalized, not requiring supplemental oxygen, but requiring ongoing medical care (COVID-19 related or otherwise), 6=Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care (used if hospitalization was extended for infection-control reasons), 7=Not hospitalized, limitation on activities, and/or requiring home oxygen, 8=Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status.
Time Frame: Baseline, Day 28
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 87 | 45
score on a scale | 3.542 (0.130) | 3.612 (0.174)

6. Secondary Outcome: Percentage of Participants With Disease Resolution at Day 14
Description: as for outcome 3
Time Frame: At Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MP1032 300mg + SoC: Participants received MP1032 300mg hard gelatin capsules orally, BID with hospital selected SoC procedure for 28 days.
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 82 | 43
percentage of participants | 84.1 [74.417 to 91.280] | 72.1 [56.331 to 84.671]

7. Secondary Outcome: All-cause Mortality Rate up to Day 14 and Day 60
Description: The percentage of participants who died by Day 14 and Day 60 were reported.
Time Frame: Up to Day 14 and Day 60
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 83 | 43
percentage of participants
  Day 14 | 1.2 [0.030 to 6.531] | 2.3 [0.059 to 12.289]
  Day 60: number analyzed (Participants) | 80 | 41
  Day 60 | 3.8 [0.780 to 10.570] | 4.9 [0.596 to 16.533]

8. Secondary Outcome: Change From Baseline in Clinical Status Score Related to COVID-19 According to the NIAID 8-point Ordinal Scale at Day 14
Description: The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status. The change from baseline in NIAID clinical status score related to COVID-19 at Day 14 were reported.
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 82 | 43
score on a scale | 2.987 (0.174) | 2.543 (0.242)

9. Secondary Outcome: Percentage of Participants Who Required Invasive Ventilation (Mechanical Ventilator and/ ECMO), or Who Died at Day 14 and Day 28
Description: Percentage of participants who required invasive mechanical ventilation/ECMO or who died by Day 14 and Day 28 were reported.
Time Frame: At Day 14 and Day 28
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 82 | 43
percentage of participants
  Day 14 | 1.2 [0.031 to 6.608] | 2.3 [0.059 to 12.289]
  Day 28: number analyzed (Participants) | 79 | 41
  Day 28 | 2.5 [0.308 to 8.848] | 2.4 [0.062 to 12.855]

10. Secondary Outcome: Change From Baseline in Clinical Status Score of the NIAID 8-point Ordinal Scale at Each Visit
Description: The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status. The change from baseline in NIAID clinical status score at each visit were reported.
Time Frame: Baseline up to Day 60
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 86 | 44
score on a scale
  Day 2 | 0.1 (0.42) | 0.0 (0.21)
  Day 3: number analyzed (Participants) | 85 | 44
  Day 3 | 0.2 (0.73) | 0.1 (0.46)
  Day 4: number analyzed (Participants) | 85 | 44
  Day 4 | 0.2 (0.83) | 0.2 (0.53)
  Day 5: number analyzed (Participants) | 84 | 44
  Day 5 | 0.4 (0.88) | 0.3 (0.70)
  Day 6: number analyzed (Participants) | 81 | 44
  Day 6 | 0.6 (1.01) | 0.4 (0.76)
  Day 7: number analyzed (Participants) | 83 | 43
  Day 7 | 1.2 (1.44) | 1.0 (1.34)
  Day 8: number analyzed (Participants) | 76 | 43
  Day 8 | 1.6 (1.60) | 1.6 (1.75)
  Day 9: number analyzed (Participants) | 75 | 39
  Day 9 | 2.0 (1.70) | 1.7 (1.77)
  Day 10: number analyzed (Participants) | 74 | 38
  Day 10 | 2.2 (1.69) | 1.7 (1.83)
  Day 11: number analyzed (Participants) | 73 | 38
  Day 11 | 2.3 (1.65) | 1.9 (1.82)
  Day 12: number analyzed (Participants) | 70 | 37
  Day 12 | 2.5 (1.66) | 1.9 (1.82)
  Day 13: number analyzed (Participants) | 68 | 34
  Day 13 | 2.7 (1.64) | 2.2 (1.71)
  Day 14: number analyzed (Participants) | 82 | 43
  Day 14 | 3.0 (1.47) | 2.6 (1.72)
  Day 28: number analyzed (Participants) | 78 | 40
  Day 28 | 3.7 (0.89) | 3.7 (0.51)
  Day 60: number analyzed (Participants) | 74 | 38
  Day 60 | 3.7 (1.01) | 3.8 (0.49)

11. Secondary Outcome: Time to (First) Improvement of at Least 1 Category on the NIAID 8-point Ordinal Scale
Description: The NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. Participants who did not improve at least 1 category on the NIAID scale or died before Day 28 were censored at Day 28. The total score range was 1 to 8 where, higher score indicates improvement in the clinical status.
Time Frame: Baseline up to Day 28
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study. As the table refers to "time to improvement', here, "Overall Number of Participants Analyzed" only signifies participants with at least 1 NIAID category of improvement at any time up to Day 28.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 81 | 40
days | 7 [7.000 to 8.000] | 7 [6.000 to 8.000]

12. Secondary Outcome: Percentage of Participants With Clinical Status Improvement of at Least 1 Category From Baseline on the NIAID 8-point Ordinal Scale at Day 14 and Day 28
Description: NIAID scale is an assessment of clinical status on a given study day and was defined as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or ECMO; 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. Higher score = improvement in clinical status. Percentage of Participants with Clinical Status Improvement of at least 1 category from baseline on the NIAID 8-point Ordinal Scale at Day 14 and Day 28 were reported.
Time Frame: Baseline, Day 14 and Day 28
Population: The ITT Set corresponded with the randomized set and included all randomized participants, irrespective of any deviation from the protocol or premature discontinuation from the study drug or withdrawal from study. Here, "Number Analyzed" signifies participants for whom NIAID data were available for Day 14 and Day 28, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 87 | 45
percentage of participants
  Day 14: number analyzed (Participants) | 82 | 43
  Day 14 | 90.2 | 86.0
  Day 28: number analyzed (Participants) | 78 | 40
  Day 28 | 98.7 | 100

13. Secondary Outcome: Time to Discharge by Day 28 and Day 60
Description: Time to discharge i.e., the total duration of participant hospitalization from baseline to discharge at Day 28 and Day 60 was reported.
Time Frame: Baseline, Day 28 and Day 60
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 83 | 42
days
  Day 28: number analyzed (Participants) | 82 | 41
  Day 28 | 9 [8.000 to 10.000] | 10 [8.000 to 13.000]
  Day 60 | 9 [8.000 to 10.000] | 10 [8.000 to 13.000]

14. Secondary Outcome: Percentage of Participants Who Were Alive and Tested Negative for COVID-19 at Day 14, Day 28, and Day 60
Description: Percentage of participants who were alive and tested negative for COVID-19 at Day 14, Day 28, and Day 60 were reported.
Time Frame: At Day 14, Day 28 and Day 60
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 76 | 39
percentage of participants
  Day 14 | 67.1 [55.374 to 77.457] | 66.7 [49.783 to 80.912]
  Day 28: number analyzed (Participants) | 69 | 38
  Day 28 | 91.3 [82.028 to 96.742] | 92.1 [78.623 to 98.341]
  Day 60: number analyzed (Participants) | 67 | 31
  Day 60 | 95.5 [87.467 to 99.067] | 93.5 [78.578 to 99.209]

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse Event (AE) was any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at screening, worsens during the study, regardless of the suspected cause of the event. TEAE was defined as any adverse event which starts or worsens at any time after initiation of study drug until the end of the follow-up period at Day 60. An SAE was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. Number of participants with TEAEs and Serious TEAEs were reported.
Time Frame: Day 1 up to Day 60
Population: The Safety Set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 86 | 45
Participants
  Participants with TEAEs | 46 | 26
  Participants with Serious TEAEs | 5 | 3

16. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Sign
Description: Vital sign parameters included of systolic and diastolic blood pressure, heart rate, respiration rate, oxygen saturation (SpO2), and body temperature. Any clinically significant change in vital signs were judged by the investigator. Number of participants with clinically significant change in vital sign values were reported.
Time Frame: Day 1 up to Day 60
Population: The Safety Set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 86 | 45
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examinations
Description: Physical examination included examination of respiratory, cardiovascular, dermatological, neurological, and gastrointestinal system. Any clinically significant abnormalities in physical examination were judged by the investigator. Number of participants with clinically significant abnormalities in physical examinations findings were reported.
Time Frame: Baseline up to Day 60
Population: The Safety Set included all randomized participants who received at least 1 dose of study drug. Here, "Overall number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 86 | 45
Participants
  Body System: Abdomen- Baseline | 0 | 1
  Body System: Abdomen- Day 8: number analyzed (Participants) | 6 | 3
  Body System: Abdomen- Day 8 | 0 | 1
  Body System: Cardiovascular- Baseline | 4 | 2
  Body System: Cardiovascular-Day 8: number analyzed (Participants) | 5 | 4
  Body System: Cardiovascular-Day 8 | 0 | 1
  Body System: Cardiovascular-Day 14: number analyzed (Participants) | 6 | 2
  Body System: Cardiovascular-Day 14 | 2 | 0
  Body System: Head, Eyes, Ears, Nose, and Throat- Baseline | 8 | 7
  Body System: Head, Eyes, Ears, Nose, and Throat- Day 8: number analyzed (Participants) | 21 | 9
  Body System: Head, Eyes, Ears, Nose, and Throat- Day 8 | 0 | 2
  Body System: Head, Eyes, Ears, Nose, and Throat- Day 14: number analyzed (Participants) | 10 | 7
  Body System: Head, Eyes, Ears, Nose, and Throat- Day 14 | 0 | 2
  Body System: Neurologic- Baseline: number analyzed (Participants) | 85 | 45
  Body System: Neurologic- Baseline | 0 | 1
  Body System: Neurologic- Day 14: number analyzed (Participants) | 3 | 1
  Body System: Neurologic- Day 14 | 0 | 1
  Body System: Other- Baseline: number analyzed (Participants) | 16 | 8
  Body System: Other- Baseline | 14 | 8
  Body System: Other- Day 8: number analyzed (Participants) | 8 | 7
  Body System: Other- Day 8 | 1 | 2
  Body System: Other- Day 14: number analyzed (Participants) | 7 | 4
  Body System: Other- Day 14 | 0 | 1
  Body System: Respiratory- Baseline | 38 | 22
  Body System: Respiratory- Day 8: number analyzed (Participants) | 45 | 22
  Body System: Respiratory- Day 8 | 4 | 2
  Body System: Respiratory- Day 14: number analyzed (Participants) | 28 | 11
  Body System: Respiratory- Day 14 | 0 | 1
  Body System: Dermatologic- Baseline: number analyzed (Participants) | 85 | 45
  Body System: Dermatologic- Baseline | 0 | 1

18. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Results
Description: Clinical laboratory tests included biochemistry, hematology and urinalysis. Any clinically significant abnormalities in clinical laboratory results were judged by the investigator. Number of participants with clinically significant abnormalities in laboratory results were reported.
Time Frame: Baseline up to Day 60
Population: The Safety Set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
Number analyzed (Participants) | 86 | 45
Participants | 23 | 22

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of MP1032
Description: Cmax of MP1032 in plasma were reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1 and Day 7
Population: The Pharmacokinetic (PK) Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose. Here, "number analyzed" signifies participants who were evaluable at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Groups:
- MP1032 300mg + SoC: Participants received MP1032 300 mg hard gelatin capsules orally, BID with hospital selected SoC procedure for 28 days.
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 4
nanograms per millilitre (ng/mL)
  Day 1 | 284.15 (170.38)
  Day 7: number analyzed (Participants) | 3
  Day 7 | 279.29 (37.85)

20. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Non-zero Concentration (AUC0-t) of MP1032
Description: AUC0-t of MP1032 in plasma were reported. Geometric mean and geometric coefficient of variation percent (CV%) was reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1 and Day 7
Population: The PK Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose. Here, "number analyzed" signifies participants who were evaluable at a specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per millilitre (h*ng/mL)
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 4
hour*nanograms per millilitre (h*ng/mL)
  Day 1 | 350.40 (42.87)
  Day 7: number analyzed (Participants) | 3
  Day 7 | 251.24 (28.72)

21. Secondary Outcome: Apparent Elimination Rate Constant (Kel) of MP1032
Description: Kel was calculated using negative of the estimated slope of the linear regression of the ln-transformed plasma concentration versus time profile in the terminal elimination phase. Kel of MP1032 in plasma were reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1
Population: The PK Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose.
Measure: Mean (Standard Deviation); unit: Per hour (1/h)
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 4
Per hour (1/h) | 0.7162 (0.8851)

22. Secondary Outcome: Apparent Body Clearance (CL/F) of MP1032
Description: Cl/F was estimated as Dose/AUC0-inf. CL/F of MP1032 in plasma was reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1
Population: The PK Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (l/h)
Groups:
- MP1032 300 mg + SoC: Participants received MP1032, 300mg hard gelatin capsules orally, BID with hospital selected SoC procedure for 28 days.
Arm/Group | MP1032 300 mg + SoC
Number analyzed (Participants) | 3
liter per hour (l/h) | 625.05 (26.09)

23. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of MP1032
Description: Vz/F was estimated as Dose/(Kel x AUC0-inf). Vz/F of MP1032 in plasma was reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 3
liter | 1494.56 (130.81)

24. Secondary Outcome: Plasma Concentration Prior to the Next Dose (Ctrough) of MP1032
Description: Ctrough of MP1032 in plasma was reported.
Time Frame: Pre-dose concentration (Day 2, Day 7, and Day 8).
Population: The PK Analysis Set included all the participants who were administered active study drug and had at least 1 post-dose evaluable plasma concentration after Day 1 dose. Here, "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 4
ng/ml
  Day 2 | 9.74 (11.27)
  Day 7 | 60.79 (121.59)
  Day 8: number analyzed (Participants) | 3
  Day 8 | 66.67 (115.48)

25. Secondary Outcome: Average Observed Plasma Concentration at Steady State of MP1032
Description: Average observed plasma concentration at steady state of MP1032 was reported.
Time Frame: Pre-dose, 0.16, 0.33, 0.5, 1, 2, 8 and 24 hours post-dose at Day 1 and Day 7
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | MP1032 300mg + SoC
Number analyzed (Participants) | 4
ng/ml
  Day 1: pre-dose | 0 (0)
  Day 1: 0.16 hours post-dose | 175.7 (322.8)
  Day 1: 0.33 hours post-dose | 200.1 (84.6)
  Day 1: 0.5 hours post-dose | 140.4 (55.3)
  Day 1: 1 hour post-dose | 64.39 (34.5)
  Day 1: 2 hours post-dose | 28.55 (145.5)
  Day 1: 8 hours post-dose | 15.48 (29.7)
  Day 1: 24 hours post-dose | 19.45 (7.5)
  Day 7: pre-dose | 243.2 (0)
  Day 7: 0.16 hours post-dose: number analyzed (Participants) | 3
  Day 7: 0.16 hours post-dose | 187.3 (53.3)
  Day 7: 0.33 hours post-dose: number analyzed (Participants) | 3
  Day 7: 0.33 hours post-dose | 281.5 (55.4)
  Day 7: 0.5 hours post-dose: number analyzed (Participants) | 3
  Day 7: 0.5 hours post-dose | 178.8 (41.1)
  Day 7: 1 hour post-dose: number analyzed (Participants) | 3
  Day 7: 1 hour post-dose | 94.42 (117.8)
  Day 7: 2 hours post-dose: number analyzed (Participants) | 3
  Day 7: 2 hours post-dose | 79.55 (155.0)
  Day 7: 8 hours post-dose: number analyzed (Participants) | 3
  Day 7: 8 hours post-dose | NA (NA) — At 8 hours geomean and CV% data was not estimated due to below limit of quantification (BLOQ).
  Day 7: 24hours post-dose: number analyzed (Participants) | 3
  Day 7: 24hours post-dose | 200.0 (0)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 60
Description: Reported AEs are TEAEs that developed, worsened, or became serious during the treatment period (time from the first dose of study treatments up to 60 days). For the overview on serious AEs, other AEs and all-Cause Mortality, data were collected and evaluated during the study for Safety Population Set only (i.e, all randomized participants who received at least 1 dose of study drug). Surgical procedures that were planned before the participant was randomized in the study are not considered AEs.
Arm/Group | MP1032 300mg + SoC | Placebo + SoC
All-Cause Mortality (participants affected / at risk) | 3/86 | 2/45
Serious Adverse Events (participants affected / at risk) | 5/86 | 3/45
Other Adverse Events (participants affected / at risk) | 46/86 | 26/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP1032 300mg + SoC (N=86) | Placebo + SoC (N=45)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP1032 300mg + SoC (N=86) | Placebo + SoC (N=45)
Alanine aminotransferase increased (Investigations) | 7 | 6
Gamma-glutamyltransferase increased (Investigations) | 4 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood glucose increased (Investigations) | 1 | 3
Blood pressure increased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2
Activated partial thromboplastin time shortened (Investigations) | 0 | 1
Blood pressure systolic increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Intestinal transit time increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1
Toxic shock syndrome (Infections and infestations) | 2 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Bradycardia (Cardiac disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Neutrophilia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 0
Blood disorder (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Cyanosis (Vascular disorders) | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0
Emotional disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT04932941/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT04932941/SAP_001.pdf